CLINICAL TRIAL: NCT01894217
Title: Pilot Study: Statin Therapy to Improve Medication Adherence
Brief Title: Statin Therapy to Improve Medication Adherence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00029836
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Hypercholesterolemia; HMG COA Reductase Inhibitor Adverse Reaction
Keywords: high cholesterol; genetic testing; medication adherence; statins; Adverse Effects; Pharmacogenetic
MeSH Terms: conditions — Hypercholesterolemia; Medication Adherence | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genetic testing (Experimental): Genetic testing and reporting for SLCO1B1*5 allele
  Interventions: Genetic: Genetic testing and reporting for SLCO1B1*5 allele

INTERVENTIONS:
Genetic: Genetic testing and reporting for SLCO1B1*5 allele — Blood test for SLCO1B1*5 allele; reporting of test results to provider and participant

SUMMARY:
The purpose of this pilot study is to examine if using genetics can improve statin adherence in patients who should be taking statins but are not because of prior side effects with statins. This study will assist physicians in making a personalized health care plan for prevention of cardiovascular disease.

DETAILED DESCRIPTION:
HMG Co-A reductase inhibitors ("statins") are commonly prescribed to lower low density lipoprotein cholesterol (LDLc) and to prevent cardiovascular disease (CVD), a leading cause of morbidity and mortality. Long-term adherence to statins in the primary care environment is challenging; consequences of statin non-adherence include higher LDLc levels, hospitalizations, costs, and death due to CVD.

Medication non-adherence is complex and multifactorial and can be associated with a number of factors including medication cost, complexity of medication regimen, poor provider-patient relationship / communication, and adverse side effects. For statins, side effects such as muscle aches, cramping, and pain (referred to broadly as statin-related myopathy) are a frequent cause of non-adherence. These symptoms are non-specific and are frequent reasons for stopping statin therapy, due to patient or provider concern about the possibility of statin-related myopathy. Many patients may be needlessly deprived of the cardiovascular benefits of long-term statin use.

A genetic risk factor for statin myopathy and subsequent non-adherence has recently been identified. In a genome-wide association study, a genetic variant (named SLCO1B1*5) was a main contributor of statin myopathy. It was demonstrated that the SLCO1B1*5 variant is not only a predictor of myopathy, but also of premature statin discontinuation. The risk with the *5 allele is statin specific: greatest with simvastatin and atorvastatin use, the least with pravastatin or rosuvastatin. Therefore, the SLCO1B1*5 variant is common, can predict myopathy, subsequent non-adherence, and due to its statin-specific effects creates a novel research paradigm for personalizing statins to an individual's genetic profile. Carriers of the SLCO1B1*5 variant may do best on rosuvastatin, pravastatin, or fluvastatin whereas non-carriers may be treated with any statin.

Specific Aims:

Aim 1: To measure the effect of genotype-guided statin prescription on patients' concerns regarding the risks of statin therapy.

Aim 2: To measure and compare the effect of genotype-guided statin prescription to non-guided therapy on statin adherence in patients who are currently not adherent to statins.

The approach for this pilot study is to recruit 100 Duke University Health System (DUHS) patients who receive care at Duke Primary Care at Pickett Road (DPC) or Center for Living (CFL) clinics that have an indication for statin therapy to reduce cardiovascular risk, but are not currently taking a statin. Consented patients will be genotyped for the SLCO1B1*5 allele at the Duke Molecular Diagnostics Laboratory. Test results will be returned first to the provider along with genotype-specific strategies to revise and/or provide a new prescription for statin therapy and next to the patient along with genotype-specific information about their personal risk of side effects on certain statin therapies. The primary outcome measures will be collected through the use of online surveys administered to patients at two time points: 1) before genetic testing and 2) 4-months after testing. Additional survey elements to address the patient's demographics, beliefs and concerns about medications, history with prescription drugs (e.g., side effects and general compliance) and overall experience with genetic testing during the study will be administered as well. It is possible that subjects will re-experience symptoms of their prior statin-intolerance when re-challenged with statins as part of this study. By avoiding certain types of statins (i.e. simvastatin and atorvastatin) in carriers of the SLCO1B1*5 genetic variant and using those statins (i.e. pravastatin and rosuvastatin) that in placebo controlled trials have no increased risk of adverse events, this risk may be less likely.

Age-, sex-, diagnosis-, and provider-matched concurrent and historical controls will be created in order to compare genetically-guided with non-genetically guided therapy

ELIGIBILITY:
Inclusion Criteria:

* Current patient (defined as seen in the last year) of the Duke Primary Care at Pickett Road or Center for Living
* Age greater than or equal to 18 years
* Provider interested in prescribing statins for cardiovascular disease prevention
* Ability to provide informed consent

Exclusion Criteria:

* Prior rhabdomyolysis, defined as CK elevation > 10 times the upper limit of normal with any statin therapy
* Prior unexplained elevation in hepatic enzymes (AST or ALT > 3 times upper limit of normal) with any statin therapy
* Use of medications known to interfere with statin metabolism or disposition
* Participation in a drug research study in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Beliefs about Medicines | Baseline and four months post genetic testing
  The Beliefs about Medicines Questionnaire (BMQ) is a validated tool and assesses patients' beliefs about their medications. Specifically, the BMQ assesses patients' perceived necessity for the prescribed medication to treat their disease as well as their concerns about adverse effects of the medication. The BMQ-specific survey will be employed as applied to 1) cholesterol lowering therapy and 2) medication therapy in general. Each question is answered with a 5-point Likert scale, ranging from 1 = strongly disagree to 5 = strongly agree. Scores obtained for individual items within the Concerns or Necessities scales are summed and total scores range from 5 to 25 (higher scores indicate stronger beliefs). Perceived concerns associated with drugs have been found to be significant predictors of poorer medication adherence.
Change in Medication adherence | baseline and four month post genotyping
  Medication adherence is assessed by the 8-item Morisky medication adherence scale (MMAS). The first 7 questions of the MMAS are scored one point for 'yes' and zero points for a 'no' response; the last question is assessed using a 5-point Likert-type responses ranging from "usually" to "all the time" (usually = 1; all the time = 5). Non-adherence is defined as a score higher than zero. For the purposes of this pilot study, the MMAS is adapted to focus on cholesterol lowering therapies.

SECONDARY OUTCOMES:
Percentage of patients who meets their National Cholesterol Education Program (NCEP) low-density lipoprotein cholesterol (LDLc)goals | Four months
  Patients who received the genetically-guided intervention will be compared to matched historical controls (2:1) and concurrent controls (2:1)
Number of new statin prescriptions written | Four months
  Patients who received the genetically-guided intervention will be compared to matched historical controls (2:1) and concurrent controls (2:1)
Patient reported medication utilization, as a surrogate for medication adherence | Four months
  Patients who received the genetically-guided intervention will be compared to matched historical controls (2:1) and concurrent controls (2:1)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Voora, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Center for Living, Durham, North Carolina
  - Duke Primary Care Clinic at Pickett Road, Durham, North Carolina